CLINICAL TRIAL: NCT03458715
Title: The Efficacy and Safety of Sodium-glucose Co-transporter 2 Inhibitor or Dipeptidyl Peptidase 4 Inhibitor Added to Premix Insulin Injection Twice Daily in Uncontrolled Type 2 Diabetes Patients
Brief Title: The Efficacy of Sodium-glucose Co-transporter 2 Inhibitor or Dipeptidyl Peptidase-4 Inhibitor in Type 2 Diabetes Patients With Premix Insulin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17MMHIS083
Record Dates: First submitted 2017-10-26; First posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2017-10

CONDITIONS: Type2 Diabetes
Keywords: SGLT2 inhibitor; DPP4 inhibitor
MeSH Terms: interventions — Sodium-Glucose Transporter 2 Inhibitors; empagliflozin; Dipeptidyl-Peptidase IV Inhibitors; Linagliptin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SGLT2 inhibitor (Empagliflozin 25 MG) (Experimental): We add SGLT2 inhibitor (Empagliflozin 25 MG, oral, once daily) to type 2 diabetes patient poorly controlled with premix insulin therapy for 6 months.
  Interventions: Drug: SGLT2 inhibitor (Empagliflozin 25 MG)
- DPP4 inhibitor (Linagliptin 5 MG) (Active Comparator): We add DPP4 inhibitor (Linagliptin 5 MG, oral, once daily) to type 2 diabetes patient poorly controlled with premix insulin therapy.for 6 months.
  Interventions: Drug: DPP4 inhibitor (Linagliptin 5 MG)

INTERVENTIONS:
Drug: SGLT2 inhibitor (Empagliflozin 25 MG) — We randomized add SGLT2 inhibitor (Empagliflozin 25 MG) or DPP4 inhibitor (Linagliptin 5 MG) to type 2 diabetes patient poorly controlled with premix insulin therapy.
  Other Names: Jardiance
  Arms: SGLT2 inhibitor (Empagliflozin 25 MG)
Drug: DPP4 inhibitor (Linagliptin 5 MG) — We randomized add SGLT2 inhibitor (Empagliflozin 25 MG) or DPP4 inhibitor (Linagliptin 5 MG) to type 2 diabetes patient poorly controlled with premix insulin therapy.
  Other Names: Trajenta
  Arms: DPP4 inhibitor (Linagliptin 5 MG)

SUMMARY:
The population of type 2 diabetes increased enormously worldwide. As disease progression, uncontrolled type 2 diabetes patients need multiple daily insulin injections, but the risk of body weight gain and hypoglycemia will increase. In recent years, the newly oral anti-hypoglycemic agents developed, such as dipeptidyl peptidase-4 inhibitors (DPP4i) and sodium-glucose co-transporter 2 inhibitors (SGLT2i). The former indirectly stimulate insulin secretion and suppress glucagon through increase incretin. The later inhibit re-absorption of blood glucose in proximal renal tubule to improve hyperglycemia. According to the guideline published in 2017 by American diabetes Associations, if patients received premix insulin injections twice daily and their glycemic control can't meet the target, increase the frequency of injection such as basal bolus would be considered. However, it is difficult for some patients and it may cause more hypoglycemia and gain of body weight. Because previous report revealed dipeptidyl peptidase-4 inhibitors or sodium-glucose co-transporter 2 inhibitors added to insulin resulted in better glycemic control, but there was no direct comparison, so we design this study to observe the efficacy of these two drugs in uncontrolled diabetes patient received twice daily insulin injections.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patient received premix insulin twice daily and HbA1c>7%
* >20 years old

Exclusion Criteria:

* Type 1 diabetes and gestational diabetes
* Diabetic ketoacidosis in previous 6 months
* Urinary tract infection in previous 6 months
* Pancreatitis in previous 6 months
* estimated GFR<45 mL/min/1.73m2
* Patient whom already received DPP4 inhibitor or SGLT2 inhibitor

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-09-21 (Estimated); Study Completion 2018-11-21 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c) | measurement at baseline, 12 week and 24 week
  change in glycated hemoglobin (HbA1c) in percentage from baseline to week 24

SECONDARY OUTCOMES:
Fasting blood glucose | measurement at baseline, 12 week and 24 week
  change in fasting blood glucose in mg/dl from baseline to week 24
Postprandial blood glucose | measurement at baseline, 12 week and 24 week
  change in postprandial blood glucose in mg/dl from baseline to week 24
Body weight | measurement at baseline, 12 week and 24 week
  change in body weight in kilogram from baseline to week 24
Hypoglycemia event | recorded at 12 week and 24 week
  documented hypoglycemia (glucose monitor <70mg/dl with hypoglycemia associated symptoms) from baseline to week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology and Metabolism, Department of Internal Medicine, Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zeng YH, Liu SC, Lee CC, Sun FJ, Liu JJ. Effect of empagliflozin versus linagliptin on body composition in Asian patients with type 2 diabetes treated with premixed insulin. Sci Rep. 2022 Oct 12;12(1):17065. doi: 10.1038/s41598-022-21486-9. PMID 36224294
- [Derived] Liu SC, Lee CC, Chuang SM, Sun FJ, Zeng YH. Comparison of efficacy and safety of empagliflozin vs linagliptin added to premixed insulin in patients with uncontrolled type 2 diabetes: A randomized, open-label study. Diabetes Metab. 2021 May;47(3):101184. doi: 10.1016/j.diabet.2020.08.001. Epub 2020 Aug 19. PMID 32827752